CLINICAL TRIAL: NCT07356310
Title: Body Composition Related Evaluation of Airway Tone and Hyper-rEactivity Using Oscillometry
Acronym: BREATH-OSC
Status: Not yet recruiting | Type: Observational
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Patrick Donohue, Assistant Professor, University of Rochester
Other Study IDs: STUDY00011306
Record Dates: First submitted 2026-01-03; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Breathing; Lung Function Decreased; Asthma (Diagnosis); Obesity
MeSH Terms: conditions — Respiratory Aspiration; Respiratory Insufficiency; Asthma; Disease; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Subjects with dyspnea referred for methacholine challenge testing: Subjects with dyspnea being evaluated for asthma who are referred for methacholine challenge testing
  Interventions: Device: Oscillometer

INTERVENTIONS:
Device: Oscillometer — The tremoFlo C-100 Airwave Oscillometry System is intended to measure respiratory system impedance using the Forced Oscillation Technique (FOT).

SUMMARY:
This study will determine if airway resistance to airflow and pressure, measured by Oscillometry, is associated with abnormal findings on methacholine challenge testing and whether these findings are associated with body habitus,

ELIGIBILITY:
Inclusion Criteria:

* Willingness to perform breathing test
* Must be able to speak and understand English
* Referred for Methacholine Challenge Test

Exclusion Criteria:

* Unable to provide consent or perform oscillometry test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Up to one hundred (100) human subjects will be recruited from the following University of Rochester locations: Mary Parkes Center for Asthma, Allergy, and Pulmonary Care, the Pulmonary Clinic at Strong Memorial Hospital, and The Pulmonary Clinic at Highland Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Oscillometer | Single measurement, approximately day 1
  The oscillometer will collect an airway impedance measurement which is made up of multiple variables.

IPD SHARING:
Plan to Share IPD: Undecided